CLINICAL TRIAL: NCT04028271
Title: Comparision of Injection Pain Caused by the 'Comfort in' Injection System Versus a Traditional Syringe for Inferior Alveolar Nerve Block Anaesthesia in Primary Teeth
Brief Title: Local Anesthesia With Needle-free Injection System
Acronym: anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinem yildirim (Other)
Responsible Party: Sponsor-Investigator, Sinem yildirim, Assistant Professor, Okan University
Organization: Okan University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018/201; Marmara universty (Other: Ethical Committe)
Record Dates: First submitted 2019-07-11; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Pediatric Anesthesia; Local Anesthesia
Keywords: needle-free injection; pain
MeSH Terms: conditions — Pain | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): local anesthesia applyed with Comfort in system
  Interventions: Device: Comfort-in injection system
- conventional injection (Active Comparator): local anesthesia applyed with conventional syringe
  Interventions: Other: conventional injection with dental needle

INTERVENTIONS:
Device: Comfort-in injection system — local anesthesia during dental treatment
  Arms: experimental
Other: conventional injection with dental needle — for local anesthesia during dental treatment
  Arms: conventional injection

SUMMARY:
The purpose of this study was to compare the pain during needle insertion and injection in mandibular molars anesthetized with either traditional syringe (control) or Comfort in System (experimental).

ELIGIBILITY:
Inclusion Criteria:

* In need of treatment of right and left molar teeth of mandible,

  * Does not have any systemic disorder,
  * High level of communication that can provide logical answers to the questions we ask
  * With parental consent,
  * Volunteers who want to participate in the research
  * 6-12 years old patients who are compatible with routine dental treatments in the pediatric clinic

Exclusion Criteria:

* No need for treatment of right and left molar teeth of mandible,
* Has a systemic condition
* Low level of communication that cannot provide reasonable answers to the questions we ask
* Without parental consent
* Do not want to participate voluntarily in the research
* Do not attend a check-in
* Patients not in the 6-12 age group

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Rating Scale (PRS) | 1 year
  The PRS measures the unpleasantness or affective dimension of a child's pain experience and is used in children aged 3-17 years old. The PRS consists of a set of cartoon faces with varying facial expressions ranging from a smile/laughter to tears, and each child is asked to select the facial expression that best represents his/her experience of discomfort. Each face has a numerical value ranging from 0 (smiling face, "no hurt") to 5 (crying/screaming face, "hurts worst").
Face, Legg, Cry, Consolability Scale (FLACC) | 1 year
  The scale comprised the following parameters: (1) Face, (2) Legs, (3) Activity, (4) Cry, and (5) Consolability. Each of the five categories is scored from 0-2, which results in a minimum total score of 0 and maximumof 10. According to this scale: 0=Relaxed and comfortable (no pain); 1-3=Mild discomfort; 4-6=Moderate pain; and 7-10=Severe discomfort or pain [Willis et al., 2003]. Behavioural parameters were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No